CLINICAL TRIAL: NCT03406078
Title: A Multicentre, Randomized, Double-Blind, Placebo Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Reducing Oral Corticosteroid Use in Adults With Oral Corticosteroid Dependent Asthma (SOURCE)
Brief Title: Study to Evaluate the Efficacy and Safety of Tezepelumab in Reducing Oral Corticosteroid Use in Adults With Oral Corticosteroid Dependent Asthma
Acronym: SOURCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00009
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to either tezepelumab or matching placebo both administered subcutaneously
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection
  Interventions: Biological: Tezepelumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Reducing Oral Corticosteroid Use in Adults with Oral Corticosteroid Dependent Asthma

DETAILED DESCRIPTION:
A Multicentre, Randomized, Double-Blind, Placebo Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Reducing Oral Corticosteroid Use in Adults with Oral Corticosteroid Dependent Asthma

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have received a physician-prescribed medium- or high-dose ICS as per GINA guideline for at least 12 months
2. Subjects must have received physician prescribed LABA and high dose ICS (total daily dose >500μg fluticasone propionate dry powder formulation equivalent) for at least 3 months. The ICS and LABA can be parts of a combination product, or given by separate inhalers.
3. Additional maintenance asthma controller medications are allowed according to standard practice of care i.e., leukotriene receptor antagonists (LTRAs), theophylline, long-acting muscarinic antagonists (LAMAs), secondary ICS and cromones. The use of these medications must be documented for at least 3 months
4. Subjects must have received OCS for the treatment of asthma for at least 6 months prior to screening and on a stable dose of between ≥ 7.5 to ≤ 30mg (prednisone or prednisolone equivalent) daily or daily equivalent for at least 1 month. The OCS dose may be administered every other day (or different doses every other day); Average dose over two days = The daily dose.
5. Morning pre-bronchodilator (BD) FEV1 must be < 80% predicted normal
6. Subjects must have evidence of asthma as documented by post-BD (albuterol/salbutatomol) reversibility of FEV1 ≥12% and ≥200 mL (15-30 min after administration of 4 puffs of albuterol/salbutamol), documented either in the previous 12 months
7. Subjects must have a history of at least 1 asthma exacerbation event within 12 months
8. Minimum 10 days compliance with the morning and evening eDiary completion and OCS,ICS,LABA as well as other asthma controller medications as captured in the eDiary during the 14 days prior to randomization
9. Documented physician-diagnosed asthma for at least 12 months

Exclusion Criteria:

1. Any clinically important pulmonary disease other than asthma (e.g. active lung infection, Chronic Obstructive Pulmonary Disease (COPD), bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   Affect the safety of the subject throughout the study Influence the findings of the study or the interpretation Impede the subject's ability to complete the entire duration of study
3. History of cancer: Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible to participate in the study provided that curative therapy was completed at least 12 months prior to visit 1.Subjects who have had other malignancies are eligible provided that curative therapy was completed at least 5 years
4. A helminth parasitic infection diagnosed within 6 months prior to screening that has not been treated with, or has failed to respond to, standard of care therapy.
5. Current smokers or subjects with smoking history ≥ 10 pack-years and subjects using vaping products, including electronic cigarettes. Former smokers with a smoking history of <10 pack years and users of vaping or e-cigarette products must have stopped for at least 6 months prior to visit 1 to be eligible.
6. History of chronic alcohol or drug abuse within 12 months
7. Tuberculosis requiring treatment within the 12 months
8. History of any known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
9. Major surgery within 8 weeks prior to visit 1 or planned surgical procedures requiring general anaesthesia or in-subject status for >1 day during the conduct of the study.
10. Clinically significant asthma exacerbation, in the opinion of the Investigator, including those requiring use of systemic corticosteroids or increase in the maintenance dose of OCS within 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (20):
  - Research Site, Bakersfield, California
  - Research Site, Newark, Delaware
  - Research Site, Kissimmee, Florida
  - Research Site, Fall River, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Altoona, Pennsylvania
  - Research Site, Homestead, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
- Argentina (7):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aire
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, San Fernando
  - Research Site, San Miguel de Tucumán
- Germany (9):
  - Research Site, Aschaffenburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Koblenz
  - Research Site, Lübeck
  - Research Site, Mainz Am Rhein
  - Research Site, München
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Wroclaw
- South Korea (2):
  - Research Site, Daegu
  - Research Site, Seoul
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Manisa
- Ukraine (4):
  - Research Site, Dnipro
  - Research Site, Kherson
  - Research Site, Lutsk
  - Research Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Menzies-Gow A, Wechsler ME, Brightling CE, Korn S, Corren J, Israel E, Chupp G, Bednarczyk A, Ponnarambil S, Caveney S, Almqvist G, Golabek M, Simonsson L, Lawson K, Bowen K, Colice G; DESTINATION study investigators. Long-term safety and efficacy of tezepelumab in people with severe, uncontrolled asthma (DESTINATION): a randomised, placebo-controlled extension study. Lancet Respir Med. 2023 May;11(5):425-438. doi: 10.1016/S2213-2600(22)00492-1. Epub 2023 Jan 23. PMID 36702146
- [Derived] Wechsler ME, Menzies-Gow A, Brightling CE, Kuna P, Korn S, Welte T, Griffiths JM, Salapa K, Hellqvist A, Almqvist G, Lal H, Kaur P, Skarby T, Colice G; SOURCE study group. Evaluation of the oral corticosteroid-sparing effect of tezepelumab in adults with oral corticosteroid-dependent asthma (SOURCE): a randomised, placebo-controlled, phase 3 study. Lancet Respir Med. 2022 Jul;10(7):650-660. doi: 10.1016/S2213-2600(21)00537-3. Epub 2022 Mar 29. PMID 35364018
- [Derived] Wechsler ME, Colice G, Griffiths JM, Almqvist G, Skarby T, Piechowiak T, Kaur P, Bowen K, Hellqvist A, Mo M, Garcia Gil E. SOURCE: a phase 3, multicentre, randomized, double-blind, placebo-controlled, parallel group trial to evaluate the efficacy and safety of tezepelumab in reducing oral corticosteroid use in adults with oral corticosteroid dependent asthma. Respir Res. 2020 Oct 13;21(1):264. doi: 10.1186/s12931-020-01503-z. PMID 33050928
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00009&attachmentIdentifier=1c64c2ac-dfb7-45d2-8049-e1f6f24c70ed&fileName=d5180c00009-csp-v4_(14-May-2020).pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00009&attachmentIdentifier=8bc47970-3cdb-4463-8948-393d1ca86f50&fileName=d5180c00009-sap-ed-3_(22-Oct-2020).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 60 centres in 7 countries. A total of 243 subjects were screened between 5MAR2018 and 27SEP2019, of which 150 were randomized and treated. 93 subjects were screen failures mainly due to exclusion criteria met and/or inclusion criteria not met. Assignment was done by Interactive Voice/Web Response System(IVRS/IWRS).
Pre-assignment Details: The screening period included a Run-in (2 weeks) and an OCS optimization phase (up to 8 weeks). At the end of period, subjects were randomized in 1:1 ratio for tezepelumab or placebo. Randomization was stratified by region (Central/Eastern Europe, Western Europe and North America, Rest of the World).
Groups:
- Tezepelumab: Tezepelumab 210 mg administered every 4 weeks subcutaneously
- Placebo: Placebo administered every 4 weeks subcutaneously
Period: Overall Study
Arm/Group | Tezepelumab | Placebo
Started | 74 | 76
Completed | 68 | 73
Not Completed | 6 | 3
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tezepelumab | Placebo | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (12.1) | 53.4 (11.9) | 53.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 45 | 94
  Male | 25 | 31 | 56
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 62 | 64 | 126
  Black or African American | 1 | 0 | 1
  Asian | 11 | 11 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Other | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 10 | 14 | 24
  Not Hispanic or Latino | 64 | 62 | 126

OUTCOME MEASURES:

1. Primary Outcome: Categorized Percent Reduction From Baseline in the Daily OCS Dose While Not Losing Asthma Control
Description: Categorized percent reduction from baseline at Week 48. Percent change from baseline is defined as {final dose-baseline dose)/baseline dose}*100, and the categories of percent change from baseline in daily OCS dose are defined as: ≥90% to ≤100% reduction, ≥75% to <90% reduction, ≥50% to <75% reduction, >0% to <50% reduction, and, no change or any increase.
Time Frame: Baseline to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  >=90% to <=100% reduction | 40 | 35
  >=75% to <90% reduction | 5 | 4
  >=50% to <75% reduction | 10 | 14
  >0% to <50% reduction | 5 | 9
  no change or any increase | 14 | 14
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Test type: Superiority; p = 0.434, Proportional odds model; Response variable: categorised % reduction from baseline in final OCS dose. Covariates in the model: treatment, region and daily OCS dose at baseline; Cumulative Odds Ratio = 1.28, 95% CI 2-sided [0.69 to 2.35]

2. Secondary Outcome: Annualised Asthma Exacerbation Rate (AAER)
Description: The annualized exacerbation rate is based on exacerbations reported by the investigator in the eCRF over 48 weeks.
Time Frame: Baseline to Week 48
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per year
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Events per year | 1.38 [0.98 to 1.95] | 2.00 [1.46 to 2.74]

3. Secondary Outcome: Proportion of Subjects With 100% Reduction From Baseline in Daily OCS Dose at Week 48
Description: Proportion (expressed as a percentage) of subjects with 100% reduction from baseline in daily OCS dose at Week 48. Percent change from baseline is defined as {(final dose-baseline dose)/baseline dose}*100.
Time Frame: Baseline to Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Percentage of participants | 54.1 | 46.1

4. Secondary Outcome: Proportion of Subjects With Daily OCS Dose ≤5 mg at Week 48
Description: Proportion (expressed as a percentage) of subjects with daily OCS dose ≤5 mg at Week 48.
Time Frame: Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Percentage of participants | 71.6 | 72.4

5. Secondary Outcome: Proportion of Subjects With ≥50% Reduction From Baseline in Daily OCS Dose at Week 48
Description: Proportion (expressed as a percentage) of subjects with ≥50% reduction from baseline in daily OCS dose at Week 48. Percent change from baseline is defined as {(final dose-baseline dose)/baseline dose}*100.
Time Frame: Baseline to Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Percentage of participants | 74.3 | 69.7

6. Secondary Outcome: Change From Baseline in Pre-bronchodilator (Pre-BD) Forced Expiratory Volume in 1 Second (FEV1)
Description: Change from baseline in pre-BD FEV1 at Week 48. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Time Frame: Baseline to Week 48
Population: Number of participants analysed presents the number of subjects with an observation at Week 48. All subjects from the Full Analysis Set with at least one change from baseline value at any post baseline visit contributes to the analyses.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 65 | 64
Litre | 0.21 (0.046) | -0.04 (0.046)

7. Secondary Outcome: Change From Baseline in Weekly Mean Daily Asthma Symptom Score Via the Daily Asthma Symptom Diary
Description: Change from baseline in Asthma Symptom Diary score at Week 48. The Asthma Symptom Diary comprises of 10 items (5 items in the morning; 5 items in the evening). Asthma symptoms during night time and daytime are recorded by the patient each morning and evening in the daily diary. A daily ASD score is the mean of the 10 items. Responses for all 10 items are required to calculate the daily ASD score; otherwise, it is treated as missing. For the 7-day average asthma symptom score, scoring is done with no imputation using the mean of at least 4 of the 7 daily ASD scores as a mean weekly item score. The 7-day average ASD score ranges from 0 to 4, where 0 indicates no asthma symptoms.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 58 | 68
Score on a scale | -0.36 (0.071) | -0.26 (0.068)

8. Secondary Outcome: Change From Baseline in Weekly Mean Rescue Medication Use
Description: Change from baseline in weekly mean rescue medication use at Week 48. Daily rescue medication use is defined as: Number of night inhaler puffs + 2 x [number of night nebulizer times] + number of daytime inhaler puffs + 2 x [number of day nebulizer times]. Each timepoint is calculated as weekly means based on daily diary data.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Weekly mean rescue medication use
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 60 | 70
Weekly mean rescue medication use | -0.85 (0.280) | -0.37 (0.268)

9. Secondary Outcome: Change From Baseline in Weekly Mean Home Peak Expiratory Flow (PEF) (Morning and Evening)
Description: Change from baseline in weekly mean morning and evening peak expiratory flow (PEF) at Week 48. Home PEF testing will be performed by the subject in the morning upon awakening and in the evening at bedtime using an electronic, hand-held spirometer. Each timepoint is calculated as weekly means using at least 4 of the 7 days of PEF data.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
L/min
  morning PEF: number analyzed (Participants) | 59 | 70
  morning PEF | 13.29 (5.653) | -9.71 (5.435)
  evening PEF: number analyzed (Participants) | 59 | 68
  evening PEF | 10.05 (5.980) | -11.37 (5.749)

10. Secondary Outcome: Change From Baseline in Weekly Mean Number of Night-time Awakening Due to Asthma
Description: Change from baseline in weekly mean number (expressed as a percentage) of night time awakenings at Week 48. Night-time awakenings percentage defined as number of nights with awakenings due to asthma and requiring rescue medication divided by number of nights with data and multiplied by 100%. At least 4 out of 7 days of data is required to calculate a weekly mean.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights with awakenings
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 59 | 70
Percentage of nights with awakenings | -15.71 (3.482) | -12.79 (3.317)

11. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 6 (ACQ-6) Score
Description: Change from baseline in ACQ-6 at Week 48. The ACQ-6 captures asthma symptoms and short-acting β2-agonist use via subject-report. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 66 | 68
Score on a scale | -0.87 (0.125) | -0.51 (0.123)

12. Secondary Outcome: Change From Baseline in Standardized Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(s)+12) Total Score
Description: Change from baseline in AQLQ(S)+12 as compared to placebo at Week 48. The AQLQ(S)+12 is a questionnaire that measures the health-related quality of life experienced by asthma subjects. The total score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. AQLQ(S)+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment).
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 66 | 67
Score on a scale | 0.94 (0.124) | 0.58 (0.123)

13. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Levels Questionnaire (EQ-5D-5L) Score
Description: Change from baseline in EQ-5D-5L at Week 48. The EQ-5D-5L questionnaire assesses 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no/slight/moderate/severe/extreme problems) that reflect increasing levels of difficulty. The EQ-5D-5L scores are converted into a single index-based value (Health State Valuation), using the UK population-based weights. The Helth State Valuation is scored between 0 to 1, where higher score indicates a better health state.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 62 | 58
Score on a scale | 0.07 (0.026) | 0.00 (0.027)

14. Secondary Outcome: Number of Participants With Asthma Specific Resource Utilizations
Description: Number of participants with asthma specific resource utilizations (e.g. unscheduled physician visits, unscheduled phone calls to physicians, use of other asthma medications) over 48 weeks.
Time Frame: Baseline to Week 48
Measure: Number; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  Hospitalisation | 5 | 10
  Emergency room visit | 4 | 7
  Unscheduled visit to specialist | 29 | 41
  Home visit | 1 | 2
  Telephone call | 26 | 43
  Ambulance transport | 0 | 1

15. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire and Classroom Impairment Questionnaire (WPAI+CIQ) Score
Description: Change from baseline in WPAI+CIQ score at Week 48. The WPAI+CIQ consists of 10 questions about how asthma and asthma related issues impact a subject's ability to work, attend classes, and perform regular daily activities.
  Work (Class) productivity loss is derived by sum of percentage of missed work (class hours) due to asthma and product of percentage of actual working hours (class) times degree of asthma affecting work (class) productivity while working. Percentage of missed work (class hours) due to asthma is calculated by number of hours missed work (class) due to asthma divided by total number of hours missed work (class) plus number of hours actually worked (in class).
  Activity impairment is the degree health affected regular activities (other than work or class) rated from 0 to 10, with 0 meaning no effect, divided by 10, and then expressed as a percentage.
Time Frame: Baseline to Week 48
Population: The work productivity loss is only applicable to subjects who were employed, which is a subset of the study population. The class productivity loss is only applicable to subjects attending school, which is a subset of the study population. No subject in Placebo arm has selected the option 'in school' on the WPAI+CIQ questionnaire at Week 48.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Percentage
  Work productivity loss: number analyzed (Participants) | 22 | 21
  Work productivity loss | -6.27 (25.30) | -9.66 (36.63)
  Class productivity loss: number analyzed (Participants) | 1 | 0
  Class productivity loss | -10.00 (0) |
  Activity impairment: number analyzed (Participants) | 59 | 59
  Activity impairment | -13.2 (29.3) | -7.8 (26.4)

16. Secondary Outcome: Change From Baseline in FENO
Description: Change from baseline in fractional exhaled nitric oxide (FeNO) at week 48.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ppb
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 58 | 57
ppb | -11.71 (2.757) | -1.40 (2.774)

17. Secondary Outcome: Change From Baseline in Peripheral Blood Eosinophils
Description: Change from baseline in blood eosinophil counts at week 48.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: cells/μL
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 63 | 67
cells/μL | -83.79 (17.078) | 33.38 (16.605)

18. Secondary Outcome: Change From Baseline From Total Serum IgE
Description: Change from baseline in total serum IgE at week 48.
Time Frame: Baseline to Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: IU/mL
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 65 | 67
IU/mL | -80.66 (36.253) | 37.77 (35.621)

19. Secondary Outcome: PK: Serum Trough Concentrations
Description: Serum trough concentrations at each scheduled visit.
Time Frame: Pre-dose samples at Baseline, Week 4, Week 12, Week 24, Week 40, Week 48, Week 60
Population: The placebo arm is not applicable since it is not the experimental product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 0
μg/mL
  Baseline: number analyzed (Participants) | 73 | 0
  Baseline | 0 (0) |
  Week 4: number analyzed (Participants) | 68 | 0
  Week 4 | 10.3298 (42.31) |
  Week 12: number analyzed (Participants) | 63 | 0
  Week 12 | 17.9626 (57.85) |
  Week 24: number analyzed (Participants) | 60 | 0
  Week 24 | 18.9210 (55.83) |
  Week 40: number analyzed (Participants) | 60 | 0
  Week 40 | 16.7095 (181.44) |
  Week 48: number analyzed (Participants) | 56 | 0
  Week 48 | 13.9224 (352.35) |
  Week 60: number analyzed (Participants) | 5 | 0
  Week 60 | 3.5591 (177.36) |

20. Secondary Outcome: Immunogenicity: Incidence of Anti-drug Antibodies (ADA)
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline. Persistently positive is defined as positive at >=2 post baseline assessments (with >=16 weeks between the first and the last positive) or positive at last post baseline assessment. Transiently positive is defined as having at least one post baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Treatment boosted ADA defined as baseline positive ADA that was boosted to a 4 fold or higher level following treatment. Treatment emergent ADA defined as sum of treatment induced ADA and treatment boosted ADA.
Time Frame: Baseline to Week 60
Measure: Number; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  ADA positive at baseline and/or post-baseline (ADA prevalence) | 3 | 2
  Any baseline ADA positive | 2 | 2
  Only baseline ADA positive | 1 | 1
  Any post-baseline ADA positive | 2 | 1
  Both baseline and at least one post-baseline ADA positive | 1 | 1
  Treatment-induced ADA positive | 1 | 0
  Treatment-boosted ADA positive | 0 | 0
  TE-ADA positive (ADA incidence) | 1 | 0
  ADA persistently positive | 1 | 1
  ADA transiently positive | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 60
Arm/Group | Tezepelumab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 12/74 | 16/76
Other Adverse Events (participants affected / at risk) | 35/74 | 48/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab (N=74) | Placebo (N=76)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
H1n1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 8 (11)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab (N=74) | Placebo (N=76)
Cataract (Eye disorders) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 5 (5)
Bronchitis (Infections and infestations) | 4 (4) | 3 (3)
Bronchitis bacterial (Infections and infestations) | 6 (14) | 7 (10)
Nasopharyngitis (Infections and infestations) | 12 (14) | 19 (29)
Oral candidiasis (Infections and infestations) | 4 (4) | 4 (5)
Sinusitis (Infections and infestations) | 1 (1) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (2)
Headache (Nervous system disorders) | 3 (3) | 8 (9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (15)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Hypertension (Vascular disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03406078/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03406078/SAP_001.pdf